CLINICAL TRIAL: NCT07039266
Title: Food Allergy Registry and Awareness Campaign in Puerto Rico
Status: Not yet recruiting | Type: Observational
Sponsor: University of Puerto Rico (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2502353537A001
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Food Allergy Proved
Keywords: Food Allergy; Allergy
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Food Allergy

SUMMARY:
Food Allergies affect 8% of children and 11% of adults, and there are increasing trends worldwide. Suffering food allergies reduces the quality of life and increases ED visits, hospitalizations, and mortality. Minorities in the United States suffer an increased food allergy burden, with higher prevalence, morbidity, and decreased use of preventive measures. Limited information is available in Puerto Rico. Moreover, advances in food allergy diagnostics, prevention, and treatment offer new hope for patients. We aim to develop a de-identified physician-diagnosed food allergy registry in Puerto Rico to characterize the food allergy population demographics, comorbidities, healthcare use, treatment, and quality of life. Our second aim is to educate patients with web-based posts to improve knowledge and awareness of food allergies.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit Puerto Rican residents aged 0 -100 years diagnosed with food allergies by board-certified allergists. A food allergy diagnosis requires a positive prick skin test or specific IgE and a history of anaphylaxis or the development of cutaneous, respiratory, cardiovascular, or vomiting within 2 hours of ingestion or a positive food challenge.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Food Allergy age 0 to 100 years
Sampling Method: Non-Probability Sample
Enrollment: 151 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Participant Questionnaire | 25 min
  Demographics Food Allergy Diagnosis Food Allergy Reactions Most Recent Food Allergy Reaction Specific Food Allergy Comorbidities Management Quality of Life Educational Component

CONTACTS AND LOCATIONS:
Overall Officials: Sylvette Nazario, MD, Principal Investigator — Universidad de Puerto Rico - Recinto de Ciencias Médicas

IPD SHARING:
Plan to Share IPD: No